CLINICAL TRIAL: NCT02735889
Title: The Effect of Different Levels of Carbonation in Drinks on Glycemic Response, Gastric Emptying, Satiety and Energy Intake
Brief Title: Fizzy Drinks Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2015/01079
Record Dates: First submitted 2016-03-13; First posted 2016-04-13 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Glycemic Response; Gastric Emptying; Satiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- No carbonation (control) (Other): No carbonation (NC, control): Potable water + sugar
  Interventions: Other: No Carbonation
- Low carbonation (Active Comparator): Low carbonation (LC): Potable water + sugar + little CO2
  Interventions: Other: Low carbonation
- High carbonation (Active Comparator): High carbonation (HC): Potable water + sugar+ high CO2
  Interventions: Other: High carbonation

INTERVENTIONS:
Other: No Carbonation — 500 ml of beverage consisting of water + 10% glucose and no carbonation
  Arms: No carbonation (control)
Other: Low carbonation — 500 ml of beverage consisting of water + 10% glucose and low carbonation
  Arms: Low carbonation
Other: High carbonation — 500 ml of beverage consisting of water + 10% glucose and high carbonation
  Arms: High carbonation

SUMMARY:
The objective of this study is to compare the effect of different levels of carbonation isocaloric beverages on glycemic response (using protocol based on standardized glycemic index testing methodology), gastric emptying and satiety. It is hypothesized that carbon dioxide will delay gastric emptying, and in turn, attenuate glycemic response and enhance satiety. The use of a non-nutrient (gas) in improving glycemic response and satiety would have important health implications for the beverage industry.

DETAILED DESCRIPTION:
15-20 healthy subjects will be recruited for the study by means of advertisements, flyers and personal communications.

A randomized, cross-over design experiment with three treatments will be carried out. Three different beverages will be prepared:- No carbonation (NC): Potable water + sugar- Low carbonation (LC): Potable water + sugar + little CO2- High carbonation (HC): Potable water + sugar+ high CO2.

The outcome measures assessed will be glycemic response, gastric emptying and satiety. Glycemic response will be measured by taking capillary blood samples (<5ul) by fingerpricking with one-time use sterilized lancets. Gastric emptying will be assessed by ultrasonography methodology developed by Okabe et al, 2015. Satiety will be measured using electronic visual analogue scales assessing hunger, fullness, desire to eat, prospective consumption and thirst. In addition, participants will be asked to rate the level of effervescence of beverage, sweetness of beverage, amount of beverage consumed, as well as how pleasant the beverage was immediately after drinking of test beverage. Feelings of bloatedness will be assessed using electronic visual analogue scales administered at 0, 15, 30, 45, 60, 90,120 min from drinking of test beverage. At the end of the test session, ad libitum lunch will be served, and the amount of food and drinks consumed will be measured (by weight difference before and after serving).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Aged between 21 - 40 years old
* BMI between 18.0-30.0 kg/m2
* Blood pressure < 140/80 mmHg
* Fasting blood glucose < 6.0mmol/L
* Fasting blood glucose < 6.0mmol/L

Exclusion Criteria:

* Are a smoker
* Have symptoms or medical history of gastrointestinal, cardiovascular, diabetes, cancer or other illnesses/diseases/conditions that could affect gastric motility and appetite
* Are on prescription medication
* Had a major medical or surgical event requiring hospitalization within the preceding 3 months.
* Are taking part in other clinical trials concurrently
* Are taking part in sports at competitive/endurance levels
* Have a score equal or greater than 3.7 for restrained eating in Dutch Eating Behaviour Questionnaire.
* Have special dietary requirements or food allergies.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose concentrations in capillary blood using Hemocue | 0, 15, 30, 45, 60, 90 and 120 min after drinking test beverage
  Capillary blood glucose will be assessed at 0, 15, 30, 45, 60, 90, 120 minutes using a Hemocue system (HemoCue Glucose 201 RT Systems)

SECONDARY OUTCOMES:
Changes in cross sectional area of antrum imaged using ultrasound | 0, 5, 10, 20, 30, 40, 50, 60, 90, 120 after drinking test beverage
  Cross sectional area of antrum will be assessed at 0, 15, 30, 45, 60, 90, 120 minutes using ultrasonography.
Satiety | 0, 15, 30, 45, 60, 90 and 120 min after drinking test beverage
  Appetite ratings will be collected at 0, 15, 30, 45, 60, 90, 120 minutes after drinking test beverage using a previously validated visual analog scales [Flint, A., A. Raben, J. E. Blundell and A. Astrup (2000). "Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies." International Journal of Obesity 24(1): 38-48]
Amount of food consumed | 2.5 hr subsequent to beverage consumption
  Ad-libitum lunch will be provided 2.5 hours after beverage consumption. The weight of the foods (g) will be taken before and after consumption, and the difference will be taken to measure the amount of food consumed (g).
Energy intake | 2.5 hr subsequent to beverage consumption
  Ad-libitum lunch will be provided 2.5 hours after beverage consumption. The energy intake will be calculated from the amount of food consumed (see Outcome 4), as well as the energy content per weight (read off from the nutritional information panel provided on the packaging) to calculate the energy intake (kcal).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No